CLINICAL TRIAL: NCT03117634
Title: An Open Label-study to Compare the Efficacy of Aflibercept Monotherapy for Polypoidal Choroidal Vasculopathy Using a Modified Intensive Treat and Extend Regime to a Fixed Dosing Regimen
Brief Title: An Open Label-study to Compare the Efficacy of Aflibercept Monotherapy for Polypoidal Choroidal Vasculopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1448/31/2017
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Age Related Macular Degeneration; Polypoidal Choroidal Vasculopathy
Keywords: anti vegf; aflibercept; treat and extend
MeSH Terms: conditions — Macular Degeneration; Polypoidal Choroidal Vasculopathy | interventions — Coal Tar; aflibercept

STUDY DESIGN:
Intervention Model Description: Prospective, 2-arm, Non-inferiority, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed dosing group (2Q8) (Active Comparator): Fixed Dosing with Aflibercept 2mg will be administered at a fixed regime at 8 week intervals through to week 52.
  Interventions: Drug: Fixed Dosing with Aflibercept 2mg
- Treat and Extend group (T&E) (Experimental): Reassessment at week 12 (month 3) by repeat examination for disease activity by OCT and indocyanine green angiography (ICGA). Subsequent treatment regime of Treat and Extend with Aflibercept 2mg will depend on disease activity at this point.
  Interventions: Drug: Treat and Extend with Aflibercept 2mg

INTERVENTIONS:
Drug: Treat and Extend with Aflibercept 2mg — Drug treatment regime which allows extension of treatment interval based on disease activity
  Other Names: T&E
  Arms: Treat and Extend group (T&E)
Drug: Fixed Dosing with Aflibercept 2mg — Fixed 8 weekly dosing regime throughout the study duration
  Other Names: 2Q8
  Arms: Fixed dosing group (2Q8)

SUMMARY:
Polypoidal choroidal neovasculopathy (PCV) is a subtype of wet age related macula degeneration (AMD) occuring more commonly in the Asian population. Besides the phenotypic differences, PCV is thought to have a lesser response to anti VEGF therapy which is the mainstay of treatment for other typical wet AMD. Recent trial data suggest that a combination with photodynamic therapy may help in the visual and anatomical outcome of PCV, and emerging evidence shows favourable outcomes the newer anti VEGF agent, aflibercept 2mg monotherapy. These trials however, have assessed aflibercept in a strict 2mg every 8 weekly regime.

In the clinical setting, a significant an unmet need in the management of PCV is a tailored treatment regime. Here we propose a treatment regimen based on disease activity for PCV with aflibercept mono therapy. A limitation of the 2q8 regime is that it is fixed and does not vary regardless of polyp closure or anatomical outcome at the first time point of assessment (month 3). We hypothesize that after the initial 3 monthly injections of aflibercept, about 50% of PCV will close and become quiescent, and in the remaining 50%, a further 3 monthly injections will increase overall polyp closure rate. After a loadings phase of either 3 or 6 months, all eyes will start on a treat and extend regime (T&E), with a minimum period of 8 weeks and a maximum of 12 weeks between treatments with 2 week increments if PCV remains quiescent. The proposed study aims to evaluate the efficacy of a modified treat and extend regime based on disease activity with aflibercept monotherapy for PCV.

DETAILED DESCRIPTION:
Age related macular degeneration (AMD) is one of the leading causes of blindness worldwide. In its exudative or wet form, choroidal neovascularization (CNV) causes an exudative maculopathy resulting in sudden loss of vision with severe effects on patients' quality of life.1,2 Intra vitreal injections of anti-vascular endothelial growth factor agents (anti-VEGF) agents have become the mainstay of treatment for AMD CNV and have been shown to have favorable outcomes in most AMD CNV subtypes.3,4 In the Asian population however, a particular subtype called polypoidal choroidal vasculopathy (PCV), which affects about 50% of exudative maculopathy, has been shown to have less favorable response to anti-VEGF therapy.5,6 The EVEREST trial, a randomized controlled trial which compares the efficacy of photodynamic therapy (PDT) with or without ranibizumab for treatment of PCV showed that PDT with or without anti VEGF improved polyp closure rate on angiographic assessment but this trial did not take into account vision as a primary end point.7 PDT appears work through its effects on choroidal vasculature, hence making it relevant to PCV which is increasingly thought to be a condition on the pachychoroid spectrum.8 PDT however, as a treatment modality presents several disadvantages. Firstly, PCV often presents as a widely distributed lesion, making it difficult to treat, with a single beam of PDT. Secondly, PDT is limited in its ability to treat lesions in the peripapillary area as there is risk of damage to the optic nerve. Thirdly, features commonly associated with PCV such as a large pigment epithelial detachment (PED) or extensive submacular hemorrhages are not usually suitable for PDT. Fourthly, there is a risk of long-term choroidal atrophy especially if repeated treatments are administered.8,9

There is emerging evidence for the use of aflibercept monotherapy in PCV. Reports range from small case series and retrospective studies to larger prospective studies. Recent data from the PLANET study showed that monotherapy of aflibercept resulted in similar letter gains in visual acuity as compared to combination treatment with PDT at 1 year. Polyp closure rate was also similar between the two groups at 38.9% with monotherapy and 44.8% with combination therapy. The VAULT and APOLLO studies suggest vision and anatomical improvements with 66-72% polyp closure in 1 year.10 These trials however, use a fixed dosing regimen (3 monthly loading doses of 2mg aflibercept followed by fixed dosing every 8 weeks (2q8) totaling 7 injections in 1 year). In addition to resolution of subretinal fluid, recent studies using the novel OCT-angiography (OCT-A) to evaluate choroidal vasculature suggests re-modelling of choroidal vasculature may also be an important therapeutic effect. We reported more prominent reduction in choroidal vessel calibre after combination treatment with PDT and bevacizumab compared to bevacizumab monotherapy. The effect of Aflibercept on choroidal vasculature has been less well studied. Some evidence however, suggested aflibercept may have more profound effect on choroidal vasculature with the reducing choroidal thickness than ranibizumab or bevacizumab.

A significant unmet need in the management of PCV with anti VEGF monotherapy is a practical way of treating patients in the real world setting that maximizes efficacy with minimal number of visits and injections. Clinical trial regimes follow a rigid treatment algorithm that aim to maximize response. In the clinical setting, these regimes are impractical in "real world" patients. Regular intensive course of treatment involves lengthy visits which include consultation time, clinical examination, retinal imaging, and often an intra vitreal injection. In clinical practice this often result in treatment fatigue and in a co-payment healthcare environment in Singapore, may also result in significant financial burden to the patient and society.

While aflibercept affords an 8 weekly treatment regime which is better than other monthly anti VEGF therapy regimes, trial regimes still do not take into account individual patients' disease patterns. This study aims to take disease activity into account to tailor treatment regimes specific for patients. In addition, it aims to provide insight into the outcomes of patients on a more clinically relevant treat and extend (T&E) regime which changes the treatment tempo in relation to disease activity.

ELIGIBILITY:
Inclusion Criteria Participant

1. Male or female study participants, age >=45 years of age at the time of informed consent.
2. Best corrected ETDRS visual acuity score <= 78 (ie 20/32 or worse)
3. Diagnosis of PCV based on ICGA

   1. Presence of intra retinal or subretinal fluid/blood at the fovea as seen on OCT
   2. Treatment naïve
4. Media clarity, pupillary dilation and individual cooperation sufficient for study procedure including fundus photography.
5. Able and willing to provide informed consent.

1.2. Exclusion Criteria Participant

1. Medical condition that, in the opinion of the investigator, would preclude participation in the study (e.g.unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
2. Participation in an investigational trial within 30 days of enrolment which involves treatment with unapproved investigational drug
3. Known allergy to any component of the study drug.
4. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110 on repeated measurements). If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
5. Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
6. Systemic anti-VEGF or pro-VEGF treatment within four months prior to randomization or anticipated use during the study.

Study Eye

1. Eye with intra retinal or subretinal fluid due to other causes than PCV
2. An ocular condition is present (other than PCV) that, in the opinion of the investigator, might affect intra or sub retinal fluid or alter visual acuity during the course of the study (e.g., diabetic macula edema (DME), vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
3. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by more than three lines (i.e., cataract would be reducing acuity to worse than 20/40 if eye was otherwise normal).
4. Any intraocular surgery within 3 months of enrollment
5. Treatment with intra vitreal corticosteroids
6. History of retinal detachment or surgery for retinal detachment
7. History of vitrectomy
8. History of macular hole
9. Evidence of vitreomacular traction that may preclude resolution of macular edema > 4 disc areas of intra/sub retinal hemorrhage
10. Aphakia
11. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis

Other Eye

1. Active intraocular inflammation
2. History of uveitis

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gemmy Cheung, Principal Investigator — SNEC
Locations (1):
- Singapore National Eye Centre, Singapore, Singpore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teo KYC, Jordan-Yu JM, Tan ACS, Yeo IYS, Mathur R, Chan CM, Wong TY, Chakravarthy U, Cheung CMG. Efficacy of a novel personalised aflibercept monotherapy regimen based on polypoidal lesion closure in participants with polypoidal choroidal vasculopathy. Br J Ophthalmol. 2022 Jul;106(7):987-993. doi: 10.1136/bjophthalmol-2020-318354. Epub 2021 Feb 11. PMID 33574033

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Personalised Group: The participants received an induction phase of treatment defined as 4 weekly intravitreal aflibercept 2mg/0.05ml at week 0, week 4 and week 8. At week 12, the participants had repeat ICGA and OCT.
  At week 12, participants in this group, in whom, polypoidal lesions had completely regressed on ICGA would enter into the treat and extend (TNE)phase. Participants with presence of polypoidal lesions (PL) on ICGA (with or without fluid on OCT) would continue three 4-weekly injections till week 24, and enter TNE phase from week 24 onwards.
- Fixed Group: The participants received an induction phase of treatment defined as 4 weekly intravitreal aflibercept 2mg/0.05ml at week 0, week 4 and week 8. At week 12, all participants had repeat ICGA and OCT.
  Participants in the fixed group went on to receive fix doses of 8-weekly aflibercept 2mn/0.05ml after the induction phase for the remaining duration of the study.
Period: Overall Study
Arm/Group | Personalised Group | Fixed Group
Started | 41; 41 eyes | 13; 13 eyes
Completed | 39; 39 eyes | 13; 13 eyes
Not Completed | 2; 2 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Fixed Group: All Study participants received an induction phase of treatment defined as 4 weekly intravitreal aflibercept 2mg/0.05ml at week 0, week 4 and week 8. At week 12, all participants had repeat ICGA and OCT.
  Participants in the fixed group went on to receive fix doses of 8-weekly aflibercept 2mn/0.05ml after the induction phase for the remaining duration of the study.
- Total: Total of all reporting groups
Arm/Group | Personalised Group | Fixed Group | Total
Number analyzed (Participants) | 39 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (9.3) | 69.3 (6.6) | 69.25 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 25 | 8 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 13 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 39 | 13 | 52
Best Corrected Visual Acuity(BCVA) [Mean (Standard Deviation); unit: ETDRS Letters (units on a scale)] — Best Corrected Visual Acuity (BCVA) defined as the mono-ocular best visual acuity in the study eye by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score after manifest refraction. More letters read correctly results in a higher letter score, which represents better visual acuity.
  ETDRS Letters (units on a scale) | 58 (14.2) | 62.8 (12.6) | 60.4 (14.3)
Central sub field thickness (CSFT) [Mean (Standard Deviation); unit: microns] — Central sub field thickness (CSFT) was defined as the objective measurement of the average thickness of the macula in the central 1 mm Early Treatment Diabetic Retinopathy Study (ETDRS) grid.
  This measure is defined by the boundaries of the retina from the inner retinal boundary at the location of the inner limiting membrane (ILM) to the outer retinal boundary at Bruch's membrane (BM).
  microns | 446.5 (181.6) | 483.2 (189.3) | 464.85 (183.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA)
Description: Mean Change in Best corrected visual acuity (BCVA) from baseline to week 52 for personalized and fixed regimen.
  it is a Non-inferiority of personalized to fixed regimen for mean change in BCVA from baseline to week 52 (Non-inferiority is considered as -5 ETDRS Letters difference )
Time Frame: From Baseline to Week 52
Population: Mean Change in Best corrected visual acuity (BCVA) from baseline to week 52 for personalized and fixed regimen.
  it is a Non-inferiority of personalized to fixed regimen for mean change in BCVA from baseline to week 52
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Personalised Group | Fixed Group
Number analyzed (Participants) | 39 | 13
Number analyzed (Eyes) | 39 | 13
ETDRS Letters | 8.1 [6.5 to 10.6] | 7.9 [5.2 to 10.4]

2. Secondary Outcome: Mean Change in Central Sub Field Thickness
Description: central sub field thickness (CSFT) was defined as the average thickness of the macula in the central 1 mm ETDRS grid. Defined as the thickness from the inner retinal boundary at the location of the inner limiting membrane (ILM) to the outer retinal boundary at Bruch's membrane (BM).
  Change in the central sub field thickness (CSFT) after the treatment was assessed , the measurement was done by optical coherence tomography (OCT). the measures were taken at baseline and week 52, the change between the two measurements ( baseline to week 52) were assessed in both groups to understand the effect of treatment on CSFT
Time Frame: From Baseline to Week 52
Population: change in the central sub field thickness (CSFT) assessed by OCT from baseline to week 52 between personalised and fixed group
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Personalised Group | Fixed Group
Number analyzed (Participants) | 39 | 13
um | -248.8 (169.9) | -164.8 (148.9)

3. Secondary Outcome: Number of Participants With Complete Polypoidal Lesion Closure
Description: This measure reports the Number of participants with complete polypoidal lesion closure defined as those showing no late leakage on Indocyanine green angiography (ICGA).
Time Frame: At Week 52
Population: number of participants with complete polypoidal lesion closure as detected on Indocyanine green angiography (ICGA) as no leakage on late ICGA stage between personalised and fixed groups
Measure: Count of Participants; unit: Participants
Arm/Group | Personalised Group | Fixed Group
Number analyzed (Participants) | 39 | 13
Participants | 21 | 5

4. Secondary Outcome: Number of Injections
Description: number of aflibercept injections administered in personalised and fixed groups
Time Frame: From Baseline to Week 52
Population: number of aflibercept injections administered in the induction phase in both groups
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Personalised Group | Fixed Group
Number analyzed (Participants) | 40 | 13
Injections | 8.2 (0.9) | 8 (0)

ADVERSE EVENTS:
Time Frame: The Adverse events (AE) and serious Adverse events (SAE) were recorded on or after the date of the administration of first study treatment, for an average of 1 year.
Description: Adverse events : Any Hospitalisation for routine treatment or monitoring of the studied indication not associated with any deterioration in condition, hospitalisation for elective or preplanned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of the study and treatment on an emergency outpatient basis for an event not fulfilling the definitions of a SAE given above and not resulting in hospital admission.
Arm/Group | Personalised Group | Fixed Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/39 | 0/13
Other Adverse Events (participants affected / at risk) | 10/39 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Personalised Group (N=39) | Fixed Group (N=13)
Cancer (Gastrointestinal disorders) | 1 | 0 — Recurrence of colorectal cancer
Ulcer (Gastrointestinal disorders) | 1 | 0 — Acute duodenal ulcer
Fall (Social circumstances) | 1 | 0 — Hospitalization due to fall
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Personalised Group (N=39) | Fixed Group (N=13)
Drop in Visual Acuity (Eye disorders) | 2 | 1 — Unrelated causality- drop in visual acuity
Stye (Extra-Ocular) (Eye disorders) | 1 | 0 — Not related and unexpected causality
Punctate epithelial erosion (Eye disorders) | 1 | 1 — Unexpected, related causality resulted in epithelial erosion
Peri-orbital Oedema (Extra-Ocular) (Eye disorders) | 1 | 0 — Unexpected not related causality resulting in peri orbital oedema
Drop in vision due to cataract (Eye disorders) | 2 | 0 — Unexpected not related causality of drop in vision due to cataract in both eyes
riased intraocular pressure (Eye disorders) | 1 | 1 — unexpected and related causality of post intravitreal treatment raised intra ocular pressure
Raised blood pressure (General disorders) | 1 | 1 — Unexpected and not related causality
Rapid Active Disease Progression (Eye disorders) | 1 | 0 — Related, Unexpected

LIMITATIONS AND CAVEATS:
More participants in the personalised group(3:1)increased the power to detect outcomes. 52 week study duration may not fully demonstrate the advantages of a TNE regimen,PL closure. Study not powered to detect the difference in PL closure at month 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contract Partners shall provide to Sponsor any proposed publication or oral presentation relating to the Study or Study Drug and Results (Publications), at least thirty days prior to the intended submission or presentation in order to allow SPONSOR to review it.

If Sponsor does not notify Contract Partner within thirty (30) days of receipt of intended Publication, Contract Partner shall be free to publish.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03117634/Prot_SAP_000.pdf